CLINICAL TRIAL: NCT02263625
Title: Regional Differences In Indication for Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: DK_03
Record Dates: First submitted 2014-09-20; First posted 2014-10-13 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Ventral Hernia
Keywords: Indication; Differences
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present study is to investigate whether there are differences in indication for ventral hernia repair and surgical approach among hernia surgeons from different geographical regions of Denmark.

DETAILED DESCRIPTION:
30 outpatient consultation will be taped and distributed among hernia surgeons in different regions of Denmark. The surgeon will then be asked to answer a questionnaire regarding the treatment and surgical technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to Køge Hospital Surg. Department with ventral hernia in December 2014

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to Køge Hospital Surg. Department with ventral hernia in December 2014
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Differences in indication for ventral hernia repair | 6 months
  Number of patients offered a ventral hernia repair after primary consultation by different hernia specialists.

SECONDARY OUTCOMES:
Differences in choice of surgical technique between surgeons | 6 months
  Which surgical approach does different surgeons offer patients with a ventral hernia

CONTACTS AND LOCATIONS:
Overall Officials: Dunja Kokotovic, MS, Principal Investigator — dept. of surgery, Køge University Hospital
Locations (1):
- Køge Sygehus, Køge, Denmark